CLINICAL TRIAL: NCT06281210
Title: Non-inferiority Study in Patients With Complete Pathological Response After Neoadjuvant Chemotherapy and Negative VABB Biopsy Undergoing RT Alone, Omitting Surgical Treatment
Brief Title: Vabb After Neoadjuvant Therapy to Avoid Surgery-pCR to Avoid Breast Surgery
Acronym: BETTY-CRASY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 2034
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; HER2-positive Breast Cancer; Neoadjuvant Chemotherapy
Keywords: Triple negative breast cancer; HER2-positive breast cancer; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omission of surgical treatment (Experimental): Omission of surgical treatment in patients with complete pathological response after neoadjuvant chemotherapy and negative VABB biopsy
  Interventions: Procedure: Omission of surgical treatment

INTERVENTIONS:
Procedure: Omission of surgical treatment — Omission of surgery in patients with pCR after neoadjuvant chemotherapy and negative VABB biopsy

SUMMARY:
This single arm study aims to evaluate the efficacy and safety of a non-surgical approach, consisting of radiotherapy (RT) alone, for patients who have achieved a complete pathological response (pCR) following neoadjuvant chemotherapy (NACT). The study design involves the histological confirmation of pCR using vacuum-assisted biopsy (VABB) or vacuum-assisted excision (VAE) guided by ultrasound. The primary objective is to demonstrate that the non-surgical, RT-only treatment and follow-up approach is not inferior to the traditional surgical approach in patients with pCR after NACT.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NACT) in breast cancer is considered the "gold standard" for the treatment of locally advanced and inoperable malignancies.

In recent years, in view of the evidence gathered, it has also become a conventional treatment alternative for patients with operable disease who are possible candidates for adjuvant chemotherapy. NACT thus aims to reduce mortality and increase surgical options, while at the same time allowing in vivo chemosensitivity testing. In view of this, NACT represents the ideal setting for clinical and translational research, which nowadays also has to address the question of future treatment options.

It is indeed a source of lively debate whether chemotherapy should be considered the only possible treatment option for the patient.

This study falls into this context, the innovative aim of which is to demonstrate histologically with the use of VABB, the complete pathological response (pCR) and to avoid surgery.

The main aim of this study is to show that a non-surgical, radiotherapy-only treatment and follow-up approach is not inferior to a surgical approach for patients who have shown complete pathological response (pCR) following neoadjuvant chemotherapy (NACT), as confirmed through histological analysis of imaging-guided sampling.

Histology will be performed by sampling 4 grams of tissue by vacuum-assisted biopsy (VABB) or vacuum-assisted excision (VAE) by ultrasound guidance (on breast marker).

The hypothesis of the study is that the VAE/VABB will be used in patients with pCR at post-NACT imaging to demonstrate the absence of disease in the previous tumour bed and, accordingly, that the use of VAE/VABB with negative histology would lead to a gold standard of treatment without surgical overtreatment.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* infiltrating breast carcinoma, non-special histotype, triple negative or HER2 +, T1-T2 N0
* single lesion
* neo-adjuvant chemotherapy treatment for at least 12 weeks according to clinical practice
* conservative surgery proposal
* M0
* tumour bed identified by breast markers placed in pre NACT by radiologist

Exclusion Criteria:

* Bilateral or multicentric tumour
* Presence of microcalcifications visualised on mammography
* Presence of associated DCIS
* Positive history of previous breast cancer
* Positive history of medical or psychiatric conditions preventing adherence to the protocol
* High risk patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  Absence of disease recurrence or progression, second primary tumor, or death

SECONDARY OUTCOMES:
Positive predictive value of MRI | 6 months
  Evaluation of the accuracy of breast MRI in predicting pCR following NACT
Contrast-Enhanced Mammography (CEM) positive predictive value | 6 months
  Evaluation of the accuracy of breast CEM in predicting pCR following NACT

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Rossi, MD, Principal Investigator — European Institute of Oncology
Locations (2):
- Italy (2):
  - Istituto di Candiolo IRCCS, Candiolo, Turin
  - European Institute of Oncology, Milan